CLINICAL TRIAL: NCT01569802
Title: A Comparison of Recall Rates Between Conventional 2d Mammography and 2d Plus 3d (Tomosynthesis) Mammography in a Screening Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rose Imaging Specialists, P.A. (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11-02
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: breast cancer screening; tomosynthesis; FFDM
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- screening

SUMMARY:
The primary aim of this study is to measure, document and compare recall rates of two-dimensional plus three dimensional (2D plus 3D) (Tomosynthesis) mammography to that of 2D mammography in a screening population. This study will compare recall rates for both non-cancer and cancer cases.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female of any race and ethnicity
* The subject is asymptomatic and presents for routine screening mammography and chooses to have a combination 2D + 3D mammogram as her standard of care.

Exclusion Criteria:

* Patient chooses standard 2D mammography over a combination 2D + 3D mammogram

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: radiology clinic screening population
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2012-01

PRIMARY OUTCOMES:
Recall Rate | up to 1 year
  measure, document and compare recall rates of two-dimensional plus three dimensional (2D plus 3D) (Tomosynthesis) mammography to that of 2D mammography in a screening population

SECONDARY OUTCOMES:
Cancer detection Rate | up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- TOPS, Houston, Texas, United States